CLINICAL TRIAL: NCT00063388
Title: A Phase II Trial of Cetuximab (C225) as Therapy for Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Study in Patients With Recurrent Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-012
Record Dates: First submitted 2003-06-25; First posted 2003-06-27 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non; Small; Cell; Lung; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cerebral Palsy; Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cetuximab 400 mg/m2 intravenously (IV) (over 120 minutes) on Day 1 of Cycle 1. followed by weekly doses of 250 mg/m2 (over 60 minutes).
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: Cetuximab — Cetuximab 400 mg/m2 intravenously (IV) (over 120 minutes) on Day 1 of Cycle 1. followed by weekly doses of 250 mg/m2 (over 60 minutes).
  Other Names: Erbitux

SUMMARY:
Determine tumor response rate and time to disease progression, survival and safety in total populations.

DETAILED DESCRIPTION:
To determine the tumor response rate and time to disease progression, survival and safety in the EGFR-positive, EGFR-negative and total populations.

ELIGIBILITY:
Inclusion Criteria

1. Subjects with recurrent or progressive NSCLC with either present or prior histologic confirmation or pathologic confirmation of NSCLC
2. Subjects receiving 1 or more prior chemotherapy regimens for the treatment of recurrent/metastatic disease, including at least 1 platinum-based combination
3. Unidimensionally measurable NSCLC
4. Subjects with tumor tissue available for EGFR assessment
5. ECOG performance status of 0 or 1
6. Subjects with asymptomatic brain metastasis were eligible; however, they must have completed radiotherapy/radiosurgery at least 3 weeks prior to enrollment and have been off steroids

Exclusion Criteria

1. Women of childbearing potential who were unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study. Male subjects must also have agreed to use effective contraception
2. Women of childbearing potential using a prohibited contraceptive method
3. Women who were pregnant or breastfeeding
4. Women with a positive pregnancy test on enrollment or prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to determine the tumor response rate for single-agent cetuximab in EGFR+ subjects. | Every 8 weeks

SECONDARY OUTCOMES:
Determine the tumor response rate in the total population and in EGFR- subjects | Every 8 weeks
Time to disease progression in the EGFR+ and total populations. | Every 8 weeks
Survival in the EGFR+ and total populations. | Every 8 weeks
Safety in the EGFR+ and total populations. | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (7):
- United States (7):
  - ImClone Investigational Site, Aventura, Florida
  - ImClone Investigational Site, Miami Beach, Florida
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, South Bend, Indiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, St Louis, Missouri